CLINICAL TRIAL: NCT02098239
Title: An Open, Multiple Dose, Single Centre Study to Determine the Antibody Response to G17DT in Patients With Advanced Pancreatic Cancer.
Brief Title: Single Centre Study to Determine the Antibody Response to G17DT in Patients With Advanced Pancreatic Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Advances Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: PC2
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Jaundice; Pancreatic Cancer
MeSH Terms: conditions — Jaundice; Pancreatic Neoplasms

ARMS (2):
- Group A (Active Comparator): Jaundiced patients with bilirubin value >80 μmol/L. Received G17DT immediately prior to biliary stenting.
  Interventions: Drug: G17DT
- Group B (Active Comparator): Patients to be treated following biliary decompression or for immediate treatment if non-jaundiced. Received G17DT 2 weeks after biliary stenting when bilirubin was <40 μmol/L.
  Interventions: Drug: G17DT

INTERVENTIONS:
Drug: G17DT
  Other Names: Polyclonal Antibody Stimulator (PAS)

SUMMARY:
The study was designed to assess the effect of jaundice on the ability of G17DT to generate antibodies before and after treatment of biliary obstruction due to advances pancreatic cancer.

DETAILED DESCRIPTION:
Jaundiced patients with advanced pancreatic cancer (either locally, advanced or metastatic) were treated with G17DT either immediately (Group A), or following biliary stenting when jaundice had resolved (Group B). Patients not jaundiced at time of presentation were to enter Group B. Patients received 3 Intramuscular injections of G17DT at weeks 0, 1, and 3. A booster injection was offered to patients who had measurable anit-G17Dt antibodies but had anti-G17DT antibodies that fell below a pre-specified threshold after week 23. Patients were evaluated until study closure ort until patient death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a pancreatic adenocarcinoma (cytologically or histologically proven), not suitable for a potentially curative resection.
* If patients were jaundiced, bilirubin had to be >80 μmol/L.
* Male or female patients over 18 years of age.
* World Health Organization (WHO) performance status of 0 to 2.
* Patients with a life expectancy of at least 8 weeks.
* Patients must have given written informed consent.

Exclusion Criteria:

* Patients undergoing a potentially curative resection.
* Jaundiced patients with a bilirubin value <80 μmol/L.
* Patients not considered fit for endoscopic or percutaneous biliary stenting.
* Patients receiving any other anti-cancer therapy.
* History of other malignant disease except non-melanomatous skin cancer or in situ carcinoma of the cervix.
* Females who were pregnant, planning to become pregnant, or who were lactating.
* Patients taking part in another study involving an investigational or licensed drug or device in the three months preceding enrolment or during this study.
* Previous G17DT treatment.
* Haematological indicators:

Haemoglobin (Hb) <10.0 g/dL. White cell count (WCC) <4.0×109/L. Platelets <100×109/L.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 1999-08; Primary Completion 2002-04 (Actual); Study Completion 2002-05

PRIMARY OUTCOMES:
Pharmacodynamic | Weeks 0, 1,3,4,6,8,12, 16+
  Gastrin-17 antibodies were measured at baseline (Week 0) and measured at each post-treatment visit.
Patient Survival | Up to week 139
  The vital status of patients was monitored throughout the study and was followed until death or the end of the study.

SECONDARY OUTCOMES:
Injection Tolerability | Up to Week 16
  Tolerability was assessed by injection site during first 16 weeks after the first injection.